CLINICAL TRIAL: NCT05336409
Title: The ELiPSE-1 Study: A Phase 1, Multicenter, Open-Label Study of CNTY-101 in Subjects With Relapsed or Refractory CD19-Positive B-Cell Malignancies
Brief Title: A Study of CNTY-101 in Participants With CD19-Positive B-Cell Malignancies
Acronym: ELiPSE-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Century Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNTY-101-111-01 (ELiPSE-1)
Record Dates: First submitted 2022-04-08; First posted 2022-04-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: R/R CD19-Positive B-Cell Malignancies; Indolent Non-Hodgkin Lymphoma; Aggressive Non-Hodgkin Lymphoma
Keywords: Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Cellular therapy; Cell therapy; CNTY-101; Century Therapeutics; Induced pluripotent stem cells; CAR-NK; NK cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Interleukin-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Escalation: Schedule A (Experimental): Lymphodepleting chemotherapy (LDC) will be followed by single dose administration of CNTY-101, alone or with supplemental human recombinant interleukin 2 (IL-2).
  Interventions: Biological: CNTY-101; Biological: IL-2; Drug: Lymphodepleting Chemotherapy
- Dose Escalation: Schedule B (Experimental): LDC will be followed by administration of CNTY-101, 3 times over 3 weeks, alone or with supplemental IL-2.
  Interventions: Biological: CNTY-101; Biological: IL-2; Drug: Lymphodepleting Chemotherapy

INTERVENTIONS:
Biological: CNTY-101 — CNTY-101 cells for intravenous (IV) infusion
Biological: IL-2 — IL-2 subcutaneous (SQ) injection
Drug: Lymphodepleting Chemotherapy — LDC as prespecified in the protocol.

SUMMARY:
ELiPSE-1 is a Phase 1, multi-center, dose-finding study to evaluate the safety, pharmacokinetics, and preliminary efficacy of CNTY-101 in participants with relapsed or refractory cluster of differentiation (CD)19-positive B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CD19-positive relapsed or refractory (R/R) B-cell Non-Hodgkin's Lymphoma (NHL).
2. Must have met the following criteria for prior treatment:

   1. Participants with aggressive NHL must have received at least 2 lines of systemic therapy (if not intended for transplant, have already undergone or be unwilling or unable to undergo chimeric antigen receptor [CAR] T-cell therapy to be eligible), or at least 3 lines of systemic therapy. Previous therapy must have included a CD20-targeted agent and an anthracycline or alkylator.
   2. Participants with follicular lymphoma (FL) must have received at least 2 lines of systemic therapy and have high-risk disease. Previous therapy must have included a CD20-targeted agent and an alkylator.
   3. Participants with marginal zone lymphoma (MZL) must have received at least 2 prior systemic therapies.
3. Measurable disease on screening evaluations.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Adequate organ function.
6. Life expectancy of ≥12 weeks.

Exclusion Criteria:

1. Any condition that confounds the ability to interpret data from the study.
2. Central nervous system (CNS)-only involvement by malignancy. (Note: participants with secondary CNS involvement are allowed.)
3. Prior allogeneic stem cell transplant.
4. Presence of clinically significant CNS pathology.
5. Other comorbid conditions defined in the protocol.
6. Use of prohibited medications within the washout period defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) as Determined by the Percentage of Participants With Dose Limiting Toxicities (DLTs) and DLTs Based on Severity | Up to 28 days
Recommended Phase 2 Regimen (RP2R) as Recommended by the Safety Review Committee (SRC) | Up to 28 days

SECONDARY OUTCOMES:
Complete Response Rate (CRR) Based on Percentage of Participants Achieving Complete Response (CR) | Up to 2 years
  CRR will be determined using Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification.
Objective Response Rate (ORR) Based on Percentage of Participants Achieving CR or Partial Response (PR) | Up to 2 years
  ORR will be determined using Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as time from first response (CR or PR) to the first documentation of progressive disease (PD) or death.
Time to Treatment Response (TTR) | Day 1 up to 2 years
  TTR is defined as time from first CNTY-101 infusion to the first documentation of response (CR or PR).
Progression-Free Survival (PFS) | Day 1 up to 2 years
  PFS is defined as time from first CNTY-101 infusion to the first documentation of PD, or death from any cause, whichever occurs first
Overall Survival (OS) | Day 1 up to 2 years
  OS is defined as time from CNTY-101 infusion to death.
Cmax: Maximum Observed Plasma Concentration for CNTY-101 | Day 1 up to 2 years
Tmax: Time to Reach the Maximum Plasma Concentration for CNTY-101 | Day 1 up to 2 years
t1/2: Terminal Disposition Phase Half-life for CNTY-101 | Day 1 up to 2 years
AUC: Area under the Concentration-time Curve for CNTY-101 | Day 1 up to 2 years
Percentage of Participants With at Least one Treatment Emergent Adverse Event (TEAE) | Day 1 up to 2 years
Percentage of Participants With Clinically Significant Laboratory Abnormalities | Day 1 up to 2 years
Time to Treatment Initiation | Enrollment to first CNTY-101 infusion (up to approximately 2 weeks)
  Time to treatment initiation is defined as the time from enrollment in the study to first CNTY-101 infusion.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California San Diego, Moores Cancer Center, San Diego, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care, Inc-Kenwood, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No